CLINICAL TRIAL: NCT01894295
Title: Assessment Vitamin D Analogues Intake Pathways on the Proteins Which Involved in Metabolic Rate in Obese Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 91-03-27-18831
Record Dates: First submitted 2013-07-03; First posted 2013-07-10 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2013-07

CONDITIONS: Obesity
Keywords: Vitamin D analogues; Resting Metabolic rate; obesity
MeSH Terms: conditions — Obesity | interventions — Corn Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- Vitamin D analogue (Experimental): 1-α hydroxyvitamin D3; dose 0.25, 0.5 and 1 microgram.
  Interventions: Dietary Supplement: Vitamin D analogue
- Placebo (Placebo Comparator): Corn oil pearl Capsules 1 gram
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Placebo — Corn oil pearl Capsules 1 gram; were given to the intervention group once a day for 8 weeks
  Other Names: corn oil capsule
  Arms: Placebo
Dietary Supplement: Vitamin D analogue — 1-α hydroxyvitamin D3 dose 0.25, 0.5 and 1 microgram were given to the intervention group once a day for 8 weeks
  Other Names: 1-α hydroxyvitamin D3
  Arms: Vitamin D analogue

SUMMARY:
The aim of this double blind clinical trial study is to investigate whether alphacalcidol treatment in obese subjects can affect the resting metabolic rate. Moreover, the investigators will evaluate the pathways of Nesfatin-1, Peroxisome proliferator-activated receptor gamma (PPARγ) and eroxisome proliferator-activated receptor- coactivator-1 α (PGC1α) protein which may lead to change in metabic rate following treatment with either alphacalcidol or placebo.

ELIGIBILITY:
Inclusion Criteria:

Age 22-52 years Body mass index equal or more than 30

Exclusion Criteria:

Acute or chronic inflammatory disease History of hypertension Alcohol or drug abuse History of any condition affecting inflammatory markers Thyroid diseases Malignancies Current smoking Diabetes mellitus Sustained hypertension Heart failure Acute or chronic infections Hepatic or renal diseases Use of PPARγ agonist drug

Ages: 22 Years to 52 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Estimated)
Dates: Start 2012-06; Primary Completion 2013-06 (Actual); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Resting Metabolic Rate | Change from baseline to 8 weeks
  Measurement by indirect calorimetry.

SECONDARY OUTCOMES:
Changes of Nesfatin-1, PPARγ and PGC1α protein levels | Change from baseline to 8 weeks
  Measurement by ELISA kit

OTHER OUTCOMES:
Change of ACS and FASN Enzymes | Change from baseline to 8 weeks
  Measurement by ELISA kit

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Jalali, PhD, Study Director — Tehran University of Medical Sciences; Khadijeh Mirzaei, MS, Principal Investigator — Tehran University of Medical Sciences
Locations (1):
- TehranUMS, Tehran, Tehran Province, Iran